CLINICAL TRIAL: NCT03781609
Title: A Motor Learning Approach to Wheelchair Propulsion Training for Manual Wheelchair Users With SCI
Brief Title: Motor Learning Approach for Manual Wheelchair Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201804133
Record Dates: First submitted 2018-11-21; First posted 2018-12-20 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Spinal Cord Injuries
Keywords: manual wheelchair; wheelchair propulsion; occupational therapy; motor learning
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Roller system group (RG) (Active Comparator): A group performing motor learning manual wheelchair propulsion repetitions on a roller system.
  Interventions: Behavioral: Roller system group (RG)
- Overground group (OG) (Active Comparator): A group performing motor learning manual wheelchair propulsion repetitions overground.
  Interventions: Behavioral: Overground group (OG)
- Placebo - Wheelchair skills group (WSG) (Placebo Comparator): A group receiving conventional manual wheelchair skills training.
  Interventions: Behavioral: Placebo - Wheelchair skills group (WSG)

INTERVENTIONS:
Behavioral: Roller system group (RG) — They will first receive the standard of care that is often used in rehabilitation: a 30 minute educational session about recommended propulsion techniques with no motor learning principles implemented. In addition, they will execute 750-1250 wheelchair propulsion repetitions on the roller system per each 1 hour session (2-3 x per week for 4-6 weeks) until they reach approximately 10,000 repetitions (10 sessions). Each session will focus on minimizing the force and frequency of pushes while using longer push strokes during propulsion.
  Arms: Roller system group (RG)
Behavioral: Overground group (OG) — They will first receive the standard of care that is often used in rehabilitation: a 30 minute educational session about recommended propulsion techniques with no motor learning principles implemented. In addition, they will execute 750-1250 wheelchair propulsion repetitions overground per each 1 hour session (2-3 x per week for 4-6 weeks) until they reach approximately 10,000 repetitions (10 sessions). Each session will focus on minimizing the force and frequency of pushes while using longer push strokes during propulsion.
  Arms: Overground group (OG)
Behavioral: Placebo - Wheelchair skills group (WSG) — They will receive the standard of care that is often used in rehabilitation: a 30 minute educational session about recommended propulsion techniques with no motor learning principles implemented.
  Arms: Placebo - Wheelchair skills group (WSG)

SUMMARY:
The overall purpose of this project is to pilot test a manual wheelchair (MWC) training program based on motor learning theory to improve wheelchair propulsion for manual wheelchair users (MWUs) with spinal cord injury (SCI).

DETAILED DESCRIPTION:
The project objective is to conduct a pilot randomized control trial (RCT) examining (1) the number of task-specific repetitions required to produce change in wheelchair propulsion techniques and (2) identifying the most conducive surface (overground or on a stationary device such as rollers) for implementing a repetition-based manual wheelchair propulsion training program. The long-term goals of this research are to minimize upper extremity pain and chronic overuse injury and to increase mobility efficiency in in persons with SCI who use MWCs for everyday mobility. The current project goal is to test the effects of a repetition-based manual wheelchair propulsion training program that emphasizes the recommended clinical practice guidelines (CPG). The expected outcome will be evidence to use in training MWUs with SCI in proper propulsion techniques in order to prevent or delay pain and chronic overuse injuries and maximize mobility through efficient wheelchair propulsion techniques. The long-term impact will be implementing evidence-based MWC propulsion training in appropriate amounts to facilitate a reduction in pain and dysfunction, a reduction in health costs, and prolonged participation in major life activities for MWUs with SCI.

Our research aims are to:

1. Compare wheelchair propulsion kinematics, kinetics, and wheelchair performance changes among three independent groups (Roller Group, Overground Group, Wheelchair Skills Group).
2. Characterize the dose-response relationship of repetition-based propulsion practice.
3. Evaluate the long-term impact of propulsion training on performance in the lived environment.

A single-blind pilot RCT will be conducted. Forty-eight individuals with SCI who use MWCs and who do not follow the recommended clinical guidelines for propulsion will be recruited. Each participant will be randomized into one of three independent groups: motor learning repetitions on a roller system (RG), motor learning repetitions overground (OG), or the placebo-controlled group receiving conventional MWC skills training (WSG). The WSG will operate as a placebo by receiving basic MWC skills training-the current standard of rehabilitation care. Participants' kinematics (video motion analysis), kinetics (SmartWheel), and wheelchair performance overground (Wheelchair Propulsion Test) will be assessed pre-intervention (Baseline), immediately following intervention (Follow-up), and three months' post-intervention (3-Month Follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 to 60 years of age
* Have a mobility limitation due to SCI, which requires the use of a manual wheelchair (MWC)
* Be able to self-propel a MWC bilaterally with their upper extremities
* Plan to use a MWC for at least 75% of activities throughout the day
* Live in the community
* Understand English at a sixth-grade level or higher
* Be able to follow multi-step instructions
* Participants must be able to provide informed consent independently
* Be able to tolerate propelling their wheelchair independently for 10 meters
* Be willing to participate in three assessments and up to 13 training sessions at the Enabling Mobility in the Community Laboratory (EMC Lab).

Exclusion Criteria:

* People will be excluded if they maneuver their MWC with their lower extremities or with only one upper extremity.
* Individuals who display the proper MWC propulsion techniques during the screening process, who already follow the CPG, or whose MWC position inhibits them from following the CPG will be excluded.
* Potential participants also will be excluded if they have bilateral incoordination due to strength inequality or neurological involvement that impairs propulsion in a steady, straight line. Specifically, if a person demonstrates upper extremity strength inequalities resulting in a 12-inch deviation from a marked pathway, he or she will be excluded.
* Other exclusionary criteria include surgeries compromising the integrity of the upper extremities or cardiovascular complications within the past year.
* Potential participants will also be excluded if upper extremity or overall bodily pain is rated 8/10 or higher per the Wong-Baker FACES Numeric Pain Scale (FACES). -In addition, potential participants will be excluded if they are currently receiving medical treatment for an acute upper extremity injury, have a Stage IV pressure injury, or are currently hospitalized.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Video Motion Capture-Hand Axle relationship Change | Baseline, Up to 4 weeks post intervention and 3-month post intervention
  Kinematic data will be collected using a 3D infrared VMC system (VICON, Centennial, CO).106 The VMC system consists of 14 Vero 2.2 digital cameras to detect the location of reflective markers, which will be attached to the participant's third metacarpal and to the wheel axle of the participant's MWC. As the participant propels through the capture volume, the VMC will record the motion of the participant's third metacarpal in relation to the wheelchair axle. Hand-axle relationship will be measured in centimeters and compared across the three testing sessions. This variable corresponds to the recommendations outlined in the CPG (bringing the hand down toward the axle during recovery [hand-axle relationship].
Video Motion Capture-Push Angle Change | Baseline, Up to 4 weeks post intervention and 3-month post intervention
  Kinematic data will be collected using a 3D infrared VMC system (VICON, Centennial, CO).106 The VMC system consists of 14 Vero 2.2 digital cameras to detect the location of reflective markers, which will be attached to the participant's third metacarpal and to the wheel axle of the participant's MWC. As the participant propels through the capture volume, the VMC will record the motion of the participant's third metacarpal in relation to the wheelchair axle. Push angle will be compared across the three testing sessions. This variable corresponds to the recommendations outlined in the CPG (use longer push strokes [push angle].
Wheelchair Propulsion Test (WPT)-Number of pushes Change | Baseline, Up to 4 weeks post intervention and 3-month post intervention
  The WPT assesses wheelchair mobility and performance of MWUs. The WPT requires MWUs to propel using a self-selected natural velocity across 10 meters of a smooth, flat surface from a static start. The number of pushes needed to complete the 10 meters,will all noted. The WPT has excellent test-retest reliability (r = .72-.96), interrater reliability (r = .80-.96), and construct validity (p < .04).14 The data collected from the WPT will assist in identifying changes of propulsion performance pre- and post-intervention and how those changes relate to the Clinical Practice Guidelines for the Preservation of upper Limb function Following Spinal Cord Injury (CPG) recommendation for minimizing the frequency of pushes while retaining the same speed.
Wheelchair Propulsion Test (WPT)-time to complete 10 meter push Change | Baseline, Up to 4 weeks post intervention and 3-month post intervention
  The WPT assesses wheelchair mobility and performance of MWUs. The WPT requires MWUs to propel using a self-selected natural velocity across 10 meters of a smooth, flat surface from a static start. Observation of the participant's propulsion pattern as well as whether their hands make contact with the pushrims, recovery, time to complete the 10 meters will be collected. The WPT has excellent test-retest reliability (r = .72-.96), interrater reliability (r = .80-.96), and construct validity (p < .04).14 The data collected from the WPT will assist in identifying changes of propulsion performance pre- and post-intervention and how those changes relate to the Clinical Practice Guidelines for the Preservation of upper Limb function Following Spinal Cord Injury (CPG) recommendation for minimizing the frequency of pushes while retaining the same speed.
Wheelchair Propulsion Test (WPT)-type of propulsion pattern comparison between time points | Baseline, Up to 4 weeks post intervention and 3-month post intervention
  The WPT assesses wheelchair mobility and performance of MWUs. The WPT requires MWUs to propel using a self-selected natural velocity across 10 meters of a smooth, flat surface from a static start. The participant's dominant propulsion pattern will be noted. The WPT has excellent test-retest reliability (r = .72-.96), interrater reliability (r = .80-.96), and construct validity (p < .04).14 The data collected from the WPT will assist in identifying changes of propulsion performance pre- and post-intervention and how those changes relate to the Clinical Practice Guidelines for the Preservation of upper Limb function Following Spinal Cord Injury (CPG) recommendation for minimizing the frequency of pushes while retaining the same speed.

SECONDARY OUTCOMES:
Outdoor Propulsion Test-Total push count | Baseline, Up to 4 weeks post intervention and 3-month post intervention
  Participants will be asked to propel their wheelchair in and around the parking lot on a fixed route. This is to assess under different environment the propulsion patterns may differ from the indoor lab environment. Total propulsion counts will be recorded and compared within and between subjects.
Outdoor Propulsion Test-# of pushes meeting clinical guidelines | Baseline, Up to 4 weeks post intervention and 3-month post intervention
  Participants will be asked to propel their wheelchair in and around the parking lot on a fixed route. This is to assess under different environment the propulsion patterns may differ from the indoor lab environment. Propulsion counts will be recorded and compared within and between subjects.
Outdoor Propulsion Test-Type of propulsion pattern | Baseline, Up to 4 weeks post intervention and 3-month post intervention
  Participants will be asked to propel their wheelchair in and around the parking lot on a fixed route. This is to assess under different environment the propulsion patterns may differ from the indoor lab environment. Propulsion patterns will be recorded and compared within and between subjects.
Outdoor Propulsion Test-Time to complete route | Baseline, Up to 4 weeks post intervention and 3-month post intervention
  Participants will be asked to propel their wheelchair in and around the parking lot on a fixed route. This is to assess under different environment the propulsion patterns may differ from the indoor lab environment. Time to complete the route will be recorded and compared within and between subjects.

OTHER OUTCOMES:
Wheelchair User's Shoulder Pain Index (WUSPI) | Baseline, Up to 4 weeks post intervention and 3-month post intervention
  A self-report measure of shoulder pain in manual wheelchair users (MWUs) during functional activities. The WUSPI consists of a 15-item questionnaire addressing shoulder pain during 15 activities within four domains: transfers, wheelchair mobility, self-care, and general activities. A 10-point visual analog scale ranging from 0 (no pain) to 10 (worst pain) is used to determine pain intensity experienced during each activity. The WUSPI score (from 0 [no pain] to 150 [worst pain] across all items) indicates the participant's level of shoulder pain during functional activities. Reliability and validity have been established by sampling long-term MWUs. The WUSPI has excellent test-retest reliability (ICC = .99),3 excellent internal consistency (α = .97),3 and moderate concurrent validity (r = -.49). Excellent convergent validity was established by correlating the WUSPI with pain intensity on a numeric rating scale (r = .77; p < .003).

CONTACTS AND LOCATIONS:
Overall Officials: Kerri A Morgan, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] National Spinal Cord Injury Statistical Center. (2016). Facts and Figures at a Glance. Birmingham, AL: University of Alabama at Birmingham.
- [Background] Cott CA. Client-centred rehabilitation: client perspectives. Disabil Rehabil. 2004 Dec 16;26(24):1411-22. doi: 10.1080/09638280400000237. PMID 15764361
- [Background] Morgan KA, Engsberg JR, Gray DB. Important wheelchair skills for new manual wheelchair users: health care professional and wheelchair user perspectives. Disabil Rehabil Assist Technol. 2017 Jan;12(1):28-38. doi: 10.3109/17483107.2015.1063015. Epub 2015 Jul 3. PMID 26138222
- [Background] Cox RJ, Amsters DI, Pershouse KJ. The need for a multidisciplinary outreach service for people with spinal cord injury living in the community. Clin Rehabil. 2001 Dec;15(6):600-6. doi: 10.1191/0269215501cr453oa. PMID 11777090
- [Background] Estores IM. The consumer's perspective and the professional literature: what do persons with spinal cord injury want? J Rehabil Res Dev. 2003 Jul-Aug;40(4 Suppl 1):93-8. doi: 10.1682/jrrd.2003.08.0093. PMID 15077653
- [Background] National Spinal Cord Injury Statistical Center. (2015). Annual Statistical Report-Complete Public Version. Birmingham, AL: University of Alabama at Birmingham.
- [Background] Kaye, H. S., Kang, T., & LaPlante, M. P. (2002). Wheelchair use in the United States [abstract]. Disability Statistics Abstract, 23, 1-4.
- [Background] LaPlante MP, Kaye HS. Demographics and trends in wheeled mobility equipment use and accessibility in the community. Assist Technol. 2010 Spring;22(1):3-17; quiz 19. doi: 10.1080/10400430903501413. PMID 20402043
- [Background] Kilkens OJ, Dallmeijer AJ, De Witte LP, Van Der Woude LH, Post MW. The Wheelchair Circuit: Construct validity and responsiveness of a test to assess manual wheelchair mobility in persons with spinal cord injury. Arch Phys Med Rehabil. 2004 Mar;85(3):424-31. doi: 10.1016/j.apmr.2003.05.006. PMID 15031828
- [Background] Kilkens OJ, Post MW, Dallmeijer AJ, van Asbeck FW, van der Woude LH. Relationship between manual wheelchair skill performance and participation of persons with spinal cord injuries 1 year after discharge from inpatient rehabilitation. J Rehabil Res Dev. 2005 May-Jun;42(3 Suppl 1):65-73. doi: 10.1682/jrrd.2004.08.0093. PMID 16195964
- [Background] Ozturk A, Ucsular FD. Effectiveness of a wheelchair skills training programme for community-living users of manual wheelchairs in Turkey: a randomized controlled trial. Clin Rehabil. 2011 May;25(5):416-24. doi: 10.1177/0269215510386979. Epub 2010 Nov 8. PMID 21059666
- [Background] Bernard, B. P., Cohen, A. L., Fine, L. J., Gjessing, C. C., & McGlothlin, J. D. (1997). Elements of ergonomics programs: A primer based on workplace evaluations of musculoskeletal disorders. US Department of Health and Human Services publication, (97-117).
- [Background] Kohn, J. P. (1998). Ergonomics Process Management: A Blueprint for Quality and Compliance. Boca Raton, FL: CRC Press.
- [Background] Boninger ML, Cooper RA, Robertson RN, Rudy TE. Wrist biomechanics during two speeds of wheelchair propulsion: an analysis using a local coordinate system. Arch Phys Med Rehabil. 1997 Apr;78(4):364-72. doi: 10.1016/s0003-9993(97)90227-6. PMID 9111455
- [Background] Hoover, A. E., Cooper, R. A., Dan, D., Dvorsnak, M., Cooper, R., Fitzgerald, S. G., & Boninger, M. L. (2003). Comparing driving habits of wheelchair users: Manual versus power. In Proceedings of the Rehabilitation Engineering and Assistive Technology Society of North America (RESNA) 26th International Conference on Technology & Disability: Research, Design, Practice, and Policy, (pp. 19-23).
- [Background] Koontz AM, Yang Y, Boninger DS, Kanaly J, Cooper RA, Boninger ML, Dieruf K, Ewer L. Investigation of the performance of an ergonomic handrim as a pain-relieving intervention for manual wheelchair users. Assist Technol. 2006 Fall;18(2):123-43; quiz 145. doi: 10.1080/10400435.2006.10131912. PMID 17236472
- [Background] Akbar M, Balean G, Brunner M, Seyler TM, Bruckner T, Munzinger J, Grieser T, Gerner HJ, Loew M. Prevalence of rotator cuff tear in paraplegic patients compared with controls. J Bone Joint Surg Am. 2010 Jan;92(1):23-30. doi: 10.2106/JBJS.H.01373. PMID 20048092
- [Background] Boninger ML, Baldwin M, Cooper RA, Koontz A, Chan L. Manual wheelchair pushrim biomechanics and axle position. Arch Phys Med Rehabil. 2000 May;81(5):608-13. doi: 10.1016/s0003-9993(00)90043-1. PMID 10807100
- [Background] Collinger JL, Impink BG, Ozawa H, Boninger ML. Effect of an intense wheelchair propulsion task on quantitative ultrasound of shoulder tendons. PM R. 2010 Oct;2(10):920-5. doi: 10.1016/j.pmrj.2010.06.007. PMID 20970761
- [Background] Davidoff G, Werner R, Waring W. Compressive mononeuropathies of the upper extremity in chronic paraplegia. Paraplegia. 1991 Jan;29(1):17-24. doi: 10.1038/sc.1991.3. PMID 2023767
- [Background] Finley MA, Rasch EK, Keyser RE, Rodgers MM. The biomechanics of wheelchair propulsion in individuals with and without upper-limb impairment. J Rehabil Res Dev. 2004 May;41(3B):385-95. doi: 10.1682/jrrd.2004.03.0385. PMID 15543456
- [Background] Gellman H, Chandler DR, Petrasek J, Sie I, Adkins R, Waters RL. Carpal tunnel syndrome in paraplegic patients. J Bone Joint Surg Am. 1988 Apr;70(4):517-9. PMID 3356717
- [Background] Koontz AM, Cooper RA, Boninger ML, Yang Y, Impink BG, van der Woude LH. A kinetic analysis of manual wheelchair propulsion during start-up on select indoor and outdoor surfaces. J Rehabil Res Dev. 2005 Jul-Aug;42(4):447-58. doi: 10.1682/jrrd.2004.08.0106. PMID 16320141
- [Background] Mercer JL, Boninger M, Koontz A, Ren D, Dyson-Hudson T, Cooper R. Shoulder joint kinetics and pathology in manual wheelchair users. Clin Biomech (Bristol). 2006 Oct;21(8):781-9. doi: 10.1016/j.clinbiomech.2006.04.010. Epub 2006 Jun 30. PMID 16808992
- [Background] Richter WM, Axelson PW. Low-impact wheelchair propulsion: achievable and acceptable. J Rehabil Res Dev. 2005 May-Jun;42(3 Suppl 1):21-33. doi: 10.1682/jrrd.2004.06.0074. PMID 16195960
- [Background] Robertson RN, Boninger ML, Cooper RA, Shimada SD. Pushrim forces and joint kinetics during wheelchair propulsion. Arch Phys Med Rehabil. 1996 Sep;77(9):856-64. doi: 10.1016/s0003-9993(96)90270-1. PMID 8822674
- [Background] Collinger JL, Boninger ML, Koontz AM, Price R, Sisto SA, Tolerico ML, Cooper RA. Shoulder biomechanics during the push phase of wheelchair propulsion: a multisite study of persons with paraplegia. Arch Phys Med Rehabil. 2008 Apr;89(4):667-76. doi: 10.1016/j.apmr.2007.09.052. PMID 18373997
- [Background] Dalyan M, Cardenas DD, Gerard B. Upper extremity pain after spinal cord injury. Spinal Cord. 1999 Mar;37(3):191-5. doi: 10.1038/sj.sc.3100802. PMID 10213328
- [Background] Nichols PJ, Norman PA, Ennis JR. Wheelchair user's shoulder? Shoulder pain in patients with spinal cord lesions. Scand J Rehabil Med. 1979;11(1):29-32. PMID 419395
- [Background] Sie IH, Waters RL, Adkins RH, Gellman H. Upper extremity pain in the postrehabilitation spinal cord injured patient. Arch Phys Med Rehabil. 1992 Jan;73(1):44-8. PMID 1729973
- [Background] Boninger ML, Cooper RA, Baldwin MA, Shimada SD, Koontz A. Wheelchair pushrim kinetics: body weight and median nerve function. Arch Phys Med Rehabil. 1999 Aug;80(8):910-5. doi: 10.1016/s0003-9993(99)90082-5. PMID 10453767
- [Background] Boninger ML, Koontz AM, Sisto SA, Dyson-Hudson TA, Chang M, Price R, Cooper RA. Pushrim biomechanics and injury prevention in spinal cord injury: recommendations based on CULP-SCI investigations. J Rehabil Res Dev. 2005 May-Jun;42(3 Suppl 1):9-19. doi: 10.1682/jrrd.2004.08.0103. PMID 16195959
- [Background] Fay BT, Boninger ML, Fitzgerald SG, Souza AL, Cooper RA, Koontz AM. Manual wheelchair pushrim dynamics in people with multiple sclerosis. Arch Phys Med Rehabil. 2004 Jun;85(6):935-42. doi: 10.1016/j.apmr.2003.08.093. PMID 15179647
- [Background] Morgan KA, Tucker SM, Klaesner JW, Engsberg JR. A motor learning approach to training wheelchair propulsion biomechanics for new manual wheelchair users: A pilot study. J Spinal Cord Med. 2017 May;40(3):304-315. doi: 10.1080/10790268.2015.1120408. Epub 2015 Dec 16. PMID 26674751
- [Background] Paralyzed Veterans of America Consortium for Spinal Cord Medicine. Preservation of upper limb function following spinal cord injury: a clinical practice guideline for health-care professionals. J Spinal Cord Med. 2005;28(5):434-70. doi: 10.1080/10790268.2005.11753844. No abstract available. PMID 16869091
- [Background] Sawatzky B, DiGiovine C, Berner T, Roesler T, Katte L. The need for updated clinical practice guidelines for preservation of upper extremities in manual wheelchair users: a position paper. Am J Phys Med Rehabil. 2015 Apr;94(4):313-24. doi: 10.1097/PHM.0000000000000203. PMID 25299526
- [Background] Boninger ML, Souza AL, Cooper RA, Fitzgerald SG, Koontz AM, Fay BT. Propulsion patterns and pushrim biomechanics in manual wheelchair propulsion. Arch Phys Med Rehabil. 2002 May;83(5):718-23. doi: 10.1053/apmr.2002.32455. PMID 11994814
- [Background] Askari S, Kirby RL, Parker K, Thompson K, O'Neill J. Wheelchair propulsion test: development and measurement properties of a new test for manual wheelchair users. Arch Phys Med Rehabil. 2013 Sep;94(9):1690-8. doi: 10.1016/j.apmr.2013.03.002. Epub 2013 Mar 14. PMID 23499781
- [Background] MacPhee AH, Kirby RL, Coolen AL, Smith C, MacLeod DA, Dupuis DJ. Wheelchair skills training program: A randomized clinical trial of wheelchair users undergoing initial rehabilitation. Arch Phys Med Rehabil. 2004 Jan;85(1):41-50. doi: 10.1016/s0003-9993(03)00364-2. PMID 14970966
- [Background] Kendall MB, Ungerer G, Dorsett P. Bridging the gap: transitional rehabilitation services for people with spinal cord injury. Disabil Rehabil. 2003 Sep 2;25(17):1008-15. doi: 10.1080/0963828031000122285. PMID 12851090
- [Background] Best KL, Miller WC, Routhier F. A description of manual wheelchair skills training curriculum in entry-to-practice occupational and physical therapy programs in Canada. Disabil Rehabil Assist Technol. 2015;10(5):401-6. doi: 10.3109/17483107.2014.907368. Epub 2014 Apr 7. PMID 24702609
- [Background] Fliess-Douer O, Vanlandewijck YC, Lubel Manor G, Van Der Woude LH. A systematic review of wheelchair skills tests for manual wheelchair users with a spinal cord injury: towards a standardized outcome measure. Clin Rehabil. 2010 Oct;24(10):867-86. doi: 10.1177/0269215510367981. Epub 2010 Jun 16. PMID 20554638
- [Background] McNevin NH, Wulf G, Carlson C. Effects of attentional focus, self-control, and dyad training on motor learning: implications for physical rehabilitation. Phys Ther. 2000 Apr;80(4):373-85. doi: 10.1093/ptj/80.4.373. PMID 10758522
- [Background] Axelson, P., Chesney, D. Y., Minkel, J., & Perr, A. (1996). The manual wheelchair training guide. Santa Cruz, CA: Pax Press.
- [Background] Kirby RL, Dupuis DJ, Macphee AH, Coolen AL, Smith C, Best KL, Newton AM, Mountain AD, Macleod DA, Bonaparte JP. The wheelchair skills test (version 2.4): measurement properties. Arch Phys Med Rehabil. 2004 May;85(5):794-804. doi: 10.1016/j.apmr.2003.07.007. PMID 15129405
- [Background] Isaacson, M. (2011). Best practices by occupational and physical therapists performing seating and mobility evaluations. Assistive Technology, 23(1), 13-21.
- [Background] Mitchell, M., Jin, B. T., Kim, A. J., Giesbrecht, E. M., Miller, W. C. (2014). METTA: A tablet-based platform for monitored at-home training as demonstrated through the EPIC Wheels Wheelchair Skills Training Program. In Proceedings of the Rehabilitation Engineering and Assistive Technology Society of North America Conference. Vancouver: University of British Columbia.
- [Background] Baddeley, A. D. & Longman, D. J. A. (1978). The influence of length and frequency of training session on the rate of learning to type. Ergonomics, 21(8), 627-635.
- [Background] Karni A. The acquisition of perceptual and motor skills: a memory system in the adult human cortex. Brain Res Cogn Brain Res. 1996 Dec;5(1-2):39-48. doi: 10.1016/s0926-6410(96)00039-0. No abstract available. PMID 9049069
- [Background] Kitago T, Krakauer JW. Motor learning principles for neurorehabilitation. Handb Clin Neurol. 2013;110:93-103. doi: 10.1016/B978-0-444-52901-5.00008-3. PMID 23312633
- [Background] Korman M, Raz N, Flash T, Karni A. Multiple shifts in the representation of a motor sequence during the acquisition of skilled performance. Proc Natl Acad Sci U S A. 2003 Oct 14;100(21):12492-7. doi: 10.1073/pnas.2035019100. Epub 2003 Oct 6. PMID 14530407
- [Background] Rice I, Gagnon D, Gallagher J, Boninger M. Hand rim wheelchair propulsion training using biomechanical real-time visual feedback based on motor learning theory principles. J Spinal Cord Med. 2010;33(1):33-42. doi: 10.1080/10790268.2010.11689672. PMID 20397442
- [Background] Rice IM, Pohlig RT, Gallagher JD, Boninger ML. Handrim wheelchair propulsion training effect on overground propulsion using biomechanical real-time visual feedback. Arch Phys Med Rehabil. 2013 Feb;94(2):256-63. doi: 10.1016/j.apmr.2012.09.014. Epub 2012 Sep 26. PMID 23022092
- [Background] Boudreau SA, Farina D, Falla D. The role of motor learning and neuroplasticity in designing rehabilitation approaches for musculoskeletal pain disorders. Man Ther. 2010 Oct;15(5):410-4. doi: 10.1016/j.math.2010.05.008. Epub 2010 Jul 7. PMID 20615749
- [Background] Dayan E, Cohen LG. Neuroplasticity subserving motor skill learning. Neuron. 2011 Nov 3;72(3):443-54. doi: 10.1016/j.neuron.2011.10.008. PMID 22078504
- [Background] Lang CE, Macdonald JR, Reisman DS, Boyd L, Jacobson Kimberley T, Schindler-Ivens SM, Hornby TG, Ross SA, Scheets PL. Observation of amounts of movement practice provided during stroke rehabilitation. Arch Phys Med Rehabil. 2009 Oct;90(10):1692-8. doi: 10.1016/j.apmr.2009.04.005. PMID 19801058
- [Background] Nudo RJ. Mechanisms for recovery of motor function following cortical damage. Curr Opin Neurobiol. 2006 Dec;16(6):638-44. doi: 10.1016/j.conb.2006.10.004. Epub 2006 Nov 3. PMID 17084614
- [Background] Karni A, Meyer G, Rey-Hipolito C, Jezzard P, Adams MM, Turner R, Ungerleider LG. The acquisition of skilled motor performance: fast and slow experience-driven changes in primary motor cortex. Proc Natl Acad Sci U S A. 1998 Feb 3;95(3):861-8. doi: 10.1073/pnas.95.3.861. PMID 9448252
- [Background] Lang CE, MacDonald JR, Gnip C. Counting repetitions: an observational study of outpatient therapy for people with hemiparesis post-stroke. J Neurol Phys Ther. 2007 Mar;31(1):3-10. doi: 10.1097/01.npt.0000260568.31746.34. PMID 17419883
- [Background] Krebs HI, Hogan N, Hening W, Adamovich SV, Poizner H. Procedural motor learning in Parkinson's disease. Exp Brain Res. 2001 Dec;141(4):425-37. doi: 10.1007/s002210100871. Epub 2001 Oct 18. PMID 11810137
- [Background] Mak MK, Hui-Chan CW. Cued task-specific training is better than exercise in improving sit-to-stand in patients with Parkinson's disease: A randomized controlled trial. Mov Disord. 2008 Mar 15;23(4):501-9. doi: 10.1002/mds.21509. PMID 18074365
- [Background] Birkenmeier RL, Prager EM, Lang CE. Translating animal doses of task-specific training to people with chronic stroke in 1-hour therapy sessions: a proof-of-concept study. Neurorehabil Neural Repair. 2010 Sep;24(7):620-35. doi: 10.1177/1545968310361957. Epub 2010 Apr 27. PMID 20424192
- [Background] Kimberley TJ, Samargia S, Moore LG, Shakya JK, Lang CE. Comparison of amounts and types of practice during rehabilitation for traumatic brain injury and stroke. J Rehabil Res Dev. 2010;47(9):851-62. doi: 10.1682/jrrd.2010.02.0019. PMID 21174250
- [Background] de Groot S, Veeger HE, Hollander AP, van der Woude LH. Influence of task complexity on mechanical efficiency and propulsion technique during learning of hand rim wheelchair propulsion. Med Eng Phys. 2005 Jan;27(1):41-9. doi: 10.1016/j.medengphy.2004.08.007. PMID 15604003
- [Background] DeGroot KK, Hollingsworth HH, Morgan KA, Morris CL, Gray DB. The influence of verbal training and visual feedback on manual wheelchair propulsion. Disabil Rehabil Assist Technol. 2009 Mar;4(2):86-94. doi: 10.1080/17483100802613685. PMID 19253097
- [Background] Rice LA, Smith I, Kelleher AR, Greenwald K, Boninger ML. Impact of a wheelchair education protocol based on practice guidelines for preservation of upper-limb function: a randomized trial. Arch Phys Med Rehabil. 2014 Jan;95(1):10-19.e11. doi: 10.1016/j.apmr.2013.06.028. Epub 2013 Jul 13. PMID 23856151
- [Background] Zwinkels M, Verschuren O, Janssen TW, Ketelaar M, Takken T; Sport-2-Stay-Fit study group; Sport-2-Stay-Fit study group. Exercise training programs to improve hand rim wheelchair propulsion capacity: a systematic review. Clin Rehabil. 2014 Sep;28(9):847-61. doi: 10.1177/0269215514525181. Epub 2014 Mar 10. PMID 24615862
- [Background] Rodgers MM, Keyser RE, Rasch EK, Gorman PH, Russell PJ. Influence of training on biomechanics of wheelchair propulsion. J Rehabil Res Dev. 2001 Sep-Oct;38(5):505-11. PMID 11732828
- [Background] de Groot S, de Bruin M, Noomen SP, van der Woude LH. Mechanical efficiency and propulsion technique after 7 weeks of low-intensity wheelchair training. Clin Biomech (Bristol). 2008 May;23(4):434-41. doi: 10.1016/j.clinbiomech.2007.11.001. Epub 2008 Feb 20. PMID 18077065
- [Background] Kotajarvi BR, Basford JR, An KN, Morrow DA, Kaufman KR. The effect of visual biofeedback on the propulsion effectiveness of experienced wheelchair users. Arch Phys Med Rehabil. 2006 Apr;87(4):510-5. doi: 10.1016/j.apmr.2005.12.033. PMID 16571390
- [Background] Klaesner J, Morgan KA, Gray DB. The development of an instrumented wheelchair propulsion testing and training device. Assist Technol. 2014 Spring;26(1):24-32. doi: 10.1080/10400435.2013.792020. PMID 24800451
- [Background] Kwarciak AM, Turner JT, Guo L, Richter WM. Comparing handrim biomechanics for treadmill and overground wheelchair propulsion. Spinal Cord. 2011 Mar;49(3):457-62. doi: 10.1038/sc.2010.149. Epub 2010 Nov 2. PMID 21042332
- [Background] Stephens CL, Engsberg JR. Comparison of overground and treadmill propulsion patterns of manual wheelchair users with tetraplegia. Disabil Rehabil Assist Technol. 2010;5(6):420-7. doi: 10.3109/17483101003793420. PMID 20441443
- [Background] DiGiovine CP, Cooper RA, Boninger ML. Dynamic calibration of a wheelchair dynamometer. J Rehabil Res Dev. 2001 Jan-Feb;38(1):41-55. PMID 11322470
- [Background] Best KL, Routhier F, Miller WC. A description of manual wheelchair skills training: current practices in Canadian rehabilitation centers. Disabil Rehabil Assist Technol. 2015;10(5):393-400. doi: 10.3109/17483107.2014.907367. Epub 2014 Apr 7. PMID 24702608
- [Background] Kilkens OJ, Post MW, Dallmeijer AJ, Seelen HA, van der Woude LH. Wheelchair skills tests: a systematic review. Clin Rehabil. 2003 Jul;17(4):418-30. doi: 10.1191/0269215503cr633oa. PMID 12785251
- [Background] Belmont PJ, Owens BD, Schoenfeld AJ. Musculoskeletal Injuries in Iraq and Afghanistan: Epidemiology and Outcomes Following a Decade of War. J Am Acad Orthop Surg. 2016 Jun;24(6):341-8. doi: 10.5435/JAAOS-D-15-00123. PMID 27115793
- [Background] Blair JA, Patzkowski JC, Schoenfeld AJ, Cross Rivera JD, Grenier ES, Lehman RA Jr, Hsu JR; Skeletal Trauma Research Consortium (STReC). Spinal column injuries among Americans in the global war on terrorism. J Bone Joint Surg Am. 2012 Sep 19;94(18):e135(1-9). doi: 10.2106/JBJS.K.00502. PMID 22992883
- [Background] Blackbourne LH. Combat damage control surgery. Crit Care Med. 2008 Jul;36(7 Suppl):S304-10. doi: 10.1097/CCM.0b013e31817e2854. PMID 18594257
- [Background] Ma VY, Chan L, Carruthers KJ. Incidence, prevalence, costs, and impact on disability of common conditions requiring rehabilitation in the United States: stroke, spinal cord injury, traumatic brain injury, multiple sclerosis, osteoarthritis, rheumatoid arthritis, limb loss, and back pain. Arch Phys Med Rehabil. 2014 May;95(5):986-995.e1. doi: 10.1016/j.apmr.2013.10.032. Epub 2014 Jan 21. PMID 24462839
- [Background] National Spinal Cord Injury Statistical Center. (2016). Spinal Cord Injury Data Sheet. Birmingham: University of Alabama at Birmingham.
- [Background] Finley MA, Rodgers MM. Prevalence and identification of shoulder pathology in athletic and nonathletic wheelchair users with shoulder pain: A pilot study. J Rehabil Res Dev. 2004 May;41(3B):395-402. doi: 10.1682/jrrd.2003.02.0022. PMID 15543457
- [Background] Fritz HA, Lysack C, Luborsky MR, Messinger SD. Long-term community reintegration: concepts, outcomes and dilemmas in the case of a military service member with a spinal cord injury. Disabil Rehabil. 2015;37(16):1501-7. doi: 10.3109/09638288.2014.967415. Epub 2014 Oct 1. PMID 25270306
- [Background] Krahn GL, Suzuki R, Horner-Johnson W. Self-rated health in persons with spinal cord injury: relationship of secondary conditions, function and health status. Qual Life Res. 2009 Jun;18(5):575-84. doi: 10.1007/s11136-009-9477-z. Epub 2009 Apr 19. PMID 19381872
- [Background] Plach HL, Sells CH. Occupational performance needs of young veterans. Am J Occup Ther. 2013 Jan-Feb;67(1):73-81. doi: 10.5014/ajot.2013.003871. PMID 23245785
- [Background] Walker KA, Morgan KA, Morris CL, DeGroot KK, Hollingsworth HH, Gray DB. Development of a community mobility skills course for people who use mobility devices. Am J Occup Ther. 2010 Jul-Aug;64(4):547-54. doi: 10.5014/ajot.2010.08117. PMID 20825125
- [Background] Goins AM, Morgan K, Stephens CL, Engsberg JR. Elbow kinematics during overground manual wheelchair propulsion in individuals with tetraplegia. Disabil Rehabil Assist Technol. 2011;6(4):312-9. doi: 10.3109/17483107.2010.528143. Epub 2010 Oct 20. PMID 20961219
- [Background] Julien MC, Morgan K, Stephens CL, Standeven J, Engsberg J. Trunk and neck kinematics during overground manual wheelchair propulsion in persons with tetraplegia. Disabil Rehabil Assist Technol. 2014 May;9(3):213-8. doi: 10.3109/17483107.2013.775362. Epub 2013 Apr 2. PMID 23548111
- [Background] Will, K., Engsberg, J. R., Foreman, M., Klaesner, J., Birkenmeier, R., & Morgan, K. A. (2015). Repetition based training for efficient propulsion in new manual wheelchair users. Journal of Physical Medicine, Rehabilitation & Disabilities, 1(001), 1-9.
- [Background] Flaherty E. Using pain-rating scales with older adults. Am J Nurs. 2008 Jun;108(6):40-7; quiz 48. doi: 10.1097/01.NAJ.0000324375.02027.9f. No abstract available. PMID 18535445
- [Background] SAS Institute Inc., Cary, NC, USA.
- [Background] Gray DB, Hollingsworth HH, Stark SL, Morgan KA. Participation survey/mobility: psychometric properties of a measure of participation for people with mobility impairments and limitations. Arch Phys Med Rehabil. 2006 Feb;87(2):189-97. doi: 10.1016/j.apmr.2005.09.014. PMID 16442971
- [Background] Curtis KA, Roach KE, Applegate EB, Amar T, Benbow CS, Genecco TD, Gualano J. Development of the Wheelchair User's Shoulder Pain Index (WUSPI). Paraplegia. 1995 May;33(5):290-3. doi: 10.1038/sc.1995.65. PMID 7630657
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Toglia J, Fitzgerald KA, O'Dell MW, Mastrogiovanni AR, Lin CD. The Mini-Mental State Examination and Montreal Cognitive Assessment in persons with mild subacute stroke: relationship to functional outcome. Arch Phys Med Rehabil. 2011 May;92(5):792-8. doi: 10.1016/j.apmr.2010.12.034. PMID 21530727
- [Background] Rushton PW, Kirby RL, Miller WC. Manual wheelchair skills: objective testing versus subjective questionnaire. Arch Phys Med Rehabil. 2012 Dec;93(12):2313-8. doi: 10.1016/j.apmr.2012.06.007. Epub 2012 Jun 21. PMID 22728701
- [Background] Lindquist NJ, Loudon PE, Magis TF, Rispin JE, Kirby RL, Manns PJ. Reliability of the performance and safety scores of the wheelchair skills test version 4.1 for manual wheelchair users. Arch Phys Med Rehabil. 2010 Nov;91(11):1752-7. doi: 10.1016/j.apmr.2010.07.226. PMID 21044722
- [Background] Mountain AD, Kirby RL, Smith C. The wheelchair skills test, version 2.4: Validity of an algorithm-based questionnaire version. Arch Phys Med Rehabil. 2004 Mar;85(3):416-23. doi: 10.1016/s0003-9993(03)00427-1. PMID 15031827
- [Background] Heinemann AW, Lai JS, Magasi S, Hammel J, Corrigan JD, Bogner JA, Whiteneck GG. Measuring participation enfranchisement. Arch Phys Med Rehabil. 2011 Apr;92(4):564-71. doi: 10.1016/j.apmr.2010.07.220. Epub 2011 Mar 2. PMID 21367395
- [Background] Stinson JN, Kavanagh T, Yamada J, Gill N, Stevens B. Systematic review of the psychometric properties, interpretability and feasibility of self-report pain intensity measures for use in clinical trials in children and adolescents. Pain. 2006 Nov;125(1-2):143-57. doi: 10.1016/j.pain.2006.05.006. Epub 2006 Jun 13. PMID 16777328
- [Background] Gagnon DH, Roy A, Verrier MC, Duclos C, Craven BC, Nadeau S. Do Performance-Based Wheelchair Propulsion Tests Detect Changes Among Manual Wheelchair Users With Spinal Cord Injury During Inpatient Rehabilitation in Quebec? Arch Phys Med Rehabil. 2016 Jul;97(7):1214-8. doi: 10.1016/j.apmr.2016.02.018. Epub 2016 Mar 15. PMID 26987621
- [Background] Pradon D, Pinsault N, Zory R, Routhier F. Could mobilty performance measures be used to evaluate wheelchair skills? J Rehabil Med. 2012 Mar;44(3):276-9. doi: 10.2340/16501977-0919. PMID 22278048
- [Background] Sawatzky B, Hers N, MacGillivray MK. Relationships between wheeling parameters and wheelchair skills in adults and children with SCI. Spinal Cord. 2015 Jul;53(7):561-4. doi: 10.1038/sc.2015.29. Epub 2015 Feb 17. PMID 25687512
- [Background] Motion Analysis Corporation. HiRes Motion Analysis Corporation System. Santa Rosa, CA.
- [Background] Cowan RE, Nash MS, Collinger JL, Koontz AM, Boninger ML. Impact of surface type, wheelchair weight, and axle position on wheelchair propulsion by novice older adults. Arch Phys Med Rehabil. 2009 Jul;90(7):1076-83. doi: 10.1016/j.apmr.2008.10.034. PMID 19577019
- [Background] Three Rivers Holdings, LLC. SmartWheel. Mesa, AZ.
- [Background] Asato KT, Cooper RA, Robertson RN, Ster JF. SMARTWheels: development and testing of a system for measuring manual wheelchair propulsion dynamics. IEEE Trans Biomed Eng. 1993 Dec;40(12):1320-4. doi: 10.1109/10.250587. PMID 8125507
- [Background] Cooper RA. SMARTWheel: From concept to clinical practice. Prosthet Orthot Int. 2009 Sep;33(3):198-209. doi: 10.1080/03093640903082126. PMID 19658010
- [Background] Lui J, MacGillivray MK, Sawatzky BJ. Test-retest reliability and minimal detectable change of the SmartWheel clinical protocol. Arch Phys Med Rehabil. 2012 Dec;93(12):2367-72. doi: 10.1016/j.apmr.2012.07.008. Epub 2012 Jul 25. PMID 22842483
- [Background] ActiGraph, LLC. GT9X Activity Monitors. Pensacola, FL.
- [Background] Bailey RR, Klaesner JW, Lang CE. An accelerometry-based methodology for assessment of real-world bilateral upper extremity activity. PLoS One. 2014 Jul 28;9(7):e103135. doi: 10.1371/journal.pone.0103135. eCollection 2014. PMID 25068258
- [Background] Garcia-Masso X, Serra-Ano P, Garcia-Raffi LM, Sanchez-Perez EA, Lopez-Pascual J, Gonzalez LM. Validation of the use of Actigraph GT3X accelerometers to estimate energy expenditure in full time manual wheelchair users with spinal cord injury. Spinal Cord. 2013 Dec;51(12):898-903. doi: 10.1038/sc.2013.85. Epub 2013 Sep 3. PMID 23999111
- [Background] Nyland J, Quigley P, Huang C, Lloyd J, Harrow J, Nelson A. Preserving transfer independence among individuals with spinal cord injury. Spinal Cord. 2000 Nov;38(11):649-57. doi: 10.1038/sj.sc.3101070. PMID 11114770
- [Background] Wulf G, McNevin N, Shea CH. The automaticity of complex motor skill learning as a function of attentional focus. Q J Exp Psychol A. 2001 Nov;54(4):1143-54. doi: 10.1080/713756012. PMID 11765737
- [Background] Wulf G, Shea C, Lewthwaite R. Motor skill learning and performance: a review of influential factors. Med Educ. 2010 Jan;44(1):75-84. doi: 10.1111/j.1365-2923.2009.03421.x. PMID 20078758
- [Background] Shea, J. B. & Morgan, R. L. (1979). Contextual interference effects on the acquisition, retention, and transfer of a motor skill. Journal of Experimental Psychology: Human Learning and Memory, 5, 179-187.
- [Background] Del Rey P, Wughalter EH, Whitehurst M. The effects of contextual interference on females with varied experience in open sport skills. Res Q Exerc Sport. 1982 Jun;53(2):108-15. doi: 10.1080/02701367.1982.10605236. No abstract available. PMID 7111849
- [Background] Hall KG, Domingues DA, Cavazos R. Contextual interference effects with skilled baseball players. Percept Mot Skills. 1994 Jun;78(3 Pt 1):835-41. doi: 10.1177/003151259407800331. PMID 8084699
- [Background] Schmidt RA, Young DE, Swinnen S, Shapiro DC. Summary knowledge of results for skill acquisition: support for the guidance hypothesis. J Exp Psychol Learn Mem Cogn. 1989 Mar;15(2):352-9. doi: 10.1037//0278-7393.15.2.352. PMID 2522520
- [Background] Gevins A, Smith ME, Leong H, McEvoy L, Whitfield S, Du R, Rush G. Monitoring working memory load during computer-based tasks with EEG pattern recognition methods. Hum Factors. 1998 Mar;40(1):79-91. doi: 10.1518/001872098779480578. PMID 9579105
- [Background] Schmidt RA, Wulf G. Continuous concurrent feedback degrades skill learning: implications for training and simulation. Hum Factors. 1997 Dec;39(4):509-25. doi: 10.1518/001872097778667979. PMID 9473972
- [Background] Goodwin JE, Eckerson JM, Voll CA Jr. Testing specificity and guidance hypotheses by manipulating relative frequency of KR scheduling in motor skill acquisition. Percept Mot Skills. 2001 Dec;93(3):819-24. doi: 10.2466/pms.2001.93.3.819. PMID 11806606
- [Background] MATLAB version 7.10.0. (2010). Natick, Massachusetts: The MathWorks Inc.
- [Background] SPSS Inc. (2012). SPSS Statistics Version 21. Chicago, IL: IBM.
- [Background] Chisholm D, Toto P, Raina K, Holm M, Rogers J. Evaluating capacity to live independently and safely in the community: Performance Assessment of Self-care Skills. Br J Occup Ther. 2014 Feb;77(2):59-63. doi: 10.4276/030802214X13916969447038. PMID 25298616